CLINICAL TRIAL: NCT02583776
Title: NEONATAL HYPOGLYCEMIA and CONTINUOUS GLUCOSE MONITORING: A RANDOMIZED CONTROLLED TRIAL IN PRETERM INFANTS
Brief Title: Continuous Glucose Monitoring and Preterm Infants
Acronym: CGM&VLBWI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Padova (Other)
Collaborators: Boston Children's Hospital (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Alfonso Galderisi, MD, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 3440/AO/15
Record Dates: First submitted 2015-10-19; First posted 2015-10-22 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Infant, Very Low Birth Weight; Neonatal Hypoglycemia
Keywords: continuous glucose monitoring (cgm); neonatal hypoglycemia; very low birth weight infants (VLBWI); preterm infants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unblinded CGM (Experimental): CGM data will be "unblinded", with Hypo/hyperglycemia alarms on. Data will be recorded from CGM every three hours and intervention to adequate glucose intake will be performed to keep glycemia in normal range (72-144mg/dl) if necessary.
  Interventions: Device: Unblinded - CGM
- Blinded CGM (Other): Hypo/hyper alarms are off. CGM data will be blinded. Glucose intake will be adequate according to 2-3 capillary glycemic tests per day.
  Interventions: Device: Blinded - CGM

INTERVENTIONS:
Device: Unblinded - CGM — Data from device will be readable and alarms on
  Arms: Unblinded CGM
Device: Blinded - CGM — Data from device will be blinded and alarms off
  Arms: Blinded CGM

SUMMARY:
Neonatal hypoglycemia is associated with brain injury and impaired neurodevelopment outcomes in very low birth weight infants (VLBWI). Glycemic monitoring is usually performed by capillary or central line sampling but does not identify up to 81% of hypoglycemic episodes in preterm newborns.

The investigators aim to assess if a continuous glucose monitor (CGM) can be used to maintain euglycemia (defined as a target value 72-144mg/dl) in VLBWI.

It will be enrolled newborns ≤32 weeks gestational age and/or of birthweight ≤1500 g, within 48 hours of life, they will be randomized in two study arms, both them will wear Dexcom G4 Platinum CGM: 1) Unblinded group (UB): glucose daily intake will be modulated according to CGM (Dexcom G4 Platinum) during the first 7 days of life, alarms for hypos/hyper will be active; 2) Blinded group (B), glucose infusion rate will be modified according to 2-3 daily capillary glucose tests, alarms for hypos will be switched off. Pain at insertion will be evaluated with the validated Premature Infant Pain Profile (PIPP) scale.

The estimated numerosity is 50 patients (25 for each arm).

DETAILED DESCRIPTION:
Background - Neonatal hypoglycemia is a common event during the first week of life and has been associated to brain injuries and poor neurodevelopment. Unfortunately it may be unrecognized for several hours from its occurrence, since it is asymptomatic/poor symptomatic in newborns (Hay WW, 2009; Cornblath, 2000; Adamkin DH, 2011; Burns et al, 2008; Wong, 2013; Duvanel et al, 1999) Despite the dramatic consequences of prolonged hypoglycemia on the neonatal brain are well known, the only tool to recognize it is represented by the capillary glycemic test performed according to risk-based protocols of Neonatal Intensive Care Units (NICUs): they consider a limited window of intervention based on 2-3 glycemic tests a day (Thomas F et al, J. Diab Science Technol. 2014).

Continuous glucose monitoring systems have offered, in the last decade, a new powerful tool to recognize more hypoglycemic events in neonates than traditional monitoring. All the works developed in neonates, to date, have been aimed to evaluate the performance of the CGM devices and have been used to record the effect of medical "intervention" in the correction of hypo or hyperglycemia (Neonatal Insulin Replacement Therapy in Europe (NIRTURE, Beardsall et al, NEJM 2008; McKinlay et al, NEJM 2015) (Harris et al J Pediatrics, 2010; Beardsall et al, Arch Dis Child Fetal Neonatal 2013). The CGM has never been used to drive medical inteventions in newborns and evaluate as independent tool to improve time-in-target for glycemia.

Previous studies demonstrated that up to 81% of the hypoglycemic episodes were not detected with blood glucose measurement (Harris et al, J Pediatrics 2010). All the published studies in neonates, to date, have used Medtronic CGM systems (Medtronic, USA). No adverse effects, associated to the implant of CGM, have been reported neither in late-preterm neither in preterm newborns.

Glycemic control in terms, and moreover, in preterm newborns still represent a challenge for physicians and the wide fluctuation (both hyperglycemia and hypoglycemia) commonly observed in such population still remains difficult to be managed with traditional blood glucose monitoring (few data/day, delay of therapeutic intervention).

Aim - The study the Investigators are going to conduct is aimed to evaluate if CGM, as driver of therapeutic decisions in preterm newborns (birthweight ≤1500g, gestational age ≤32 weeks) during the first week of life, may be able to maintain "euglycemia". Euglycemia will be defined as values within the range 72-144mg/dl (4-8mmol/L)(Harris et al J Pediatrics, 2010; Beardsall et al, Arch Dis Child Fetal Neonatal Ed 2013)

Study design - Randomized Controlled Trial

* Patients: newborns with GA ≤32weeks and/or BW≤ 1500 g. They will be enrolled within the first 48 hours of life
* Intevention group: Unblinded CGM (DexcomG4Platinum) data to adequate daily glucose intake
* Control group: Blinded CGM with daily glucose intake adequated according to SMBG (=2 blood glucose/day)
* Primary Outcome: to evaluate if Unblinded CGM increases the time within "euglycemic" range (72-144mg/dl)

Materials and Methods - Dexcom G4 Platinum (Dexcom Inc, CA - USA) sensor will be applied within 48 hours from birth to the study population on the lateral side of thigh, after parents' consent collection.

All the patients will be randomized to the blinded or unblinded group before the application of CGM. Randomization will be performed using a randomization list electronically generated.

Unblinded group (intervention/open CGM group): they will wear CGM for 7 days, the alarms of CGM will be switched on and the daily intake of carbohydrates will be adapted according to CGM data. The study staff will record data every three hours in absence of hypo alarms (see below for carbs adjustment procedure).

Blinded group: they will wear CGM for 7 days, the alarms and the CGM monitor will be blinded. At least two calibrations a day, according to manufacturer instruction, will be inserted. The daily amount of carbohydrates will be decided according to blood glucose test (at least 2/day) and to recommendation of American Academy of Pediatrics (see below).

Numerosity: the estimated numerosity is 50 patients according to primary outcome. Unfortunately no data are available on this population; 10 extra patients will be recruited in case of premature interruption of recording (due to sensor detachment, malfunction, loss of the patient or interruption of monitoring due to local/systemic complication) in order to ensure a total amount of 250 days of monitoring (50% in the UB-CGM group and 50% in the B-CGM group) with a maximum amount of 350 days of monitoring. So the estimated time of monitoring is expected to be min 250, max 350 days, divided into the two groups.

Reasons for study interruption: local and/or systemic complication due to the application of device, transfer of patient to another center of care, withdrawal of consent, death, malfunction of device. Reasons for interruption of monitoring will be specified in the final report.

Carbohydrates adjustment procedure: the procedure for carbohydrates adjustment uses a worksheet described in Agus MSD, Steil G et al NEJM 2012 and adapted to NICU standard of nutrition suggested from American Academy of Pediatrics. The worksheet has been set up according to the NICU protocols in agreement with recommendation of American Academy of Pediatrics, Committee on Nutrition.

The 1st day intake is set on 6-8gr/kg of carbohydrates; a default daily increase of 1gr/kg/day in case of euglycemia is applied; such increase may variate according to the CGM data in the unblinded group or to the 2 glycemic tests performed in the blinded group in order to achieve the target as following:

i. if the average was >= 180 mg/dL decrease the calculated GIR by 1 g/kg/d ii. If the average was between 144 and 179 mg/dL do not make any adjustment iii. If the average was between 72 and 143 mg/dL check if the minimum GIR has been reached and if not increase the value to the minimum GIR for that day iv. If the average was lower than 72 mg/dL increase the rate to the either the minimum rate + 2 or the calculated rate plus 2, whichever is bigger; v. if glycemia <41mg/gl: increase of 2.8g/kg/die the GIR and perform a bolus of 2ml/kg/d of G10%.

Details of the worksheet have been described in Agus et al (NEJM2012).

Worksheet has been designed considering as follows:

Target 108,00 Low limit 72,00 High limit 144,00 Hyper Theshold 180,00 Hypo Threshold 40,00 A decrease has been considered above hyper threshold of 1g/kg/d up to a minimum GIR of 4.5g/k/d. No increase will be performed between 144 and 180mg/dl.

Data analysis will be performed as intention to treat (ITT).

Discussion: perspective and limits - Euglycemia definition remains controversial in neonatology. Even though, in our study, we have decided to adopt the NIRTURE targets (Beardsall et al, 2010) considering optimal a range from 72 mg/dl (4 mmol/L) to 144mg/dl (8 mmol/L). Values below 40mg/dl will require a G10% bolus (2ml/kg) and an increase of 2.8gr/kg of intake of carbs; values between 40 and 77mg/dl require an increase of carbs adapted to reach the middle point of the expected target. Similarly for values above the upper limit we have considered a decrease of carbs intake (minimum 4.5gr/kg/day).

The main difference between the two study groups is represented by the number of information available for the physician and, consequently, from the number of changes in glucose intake.

The use of a worksheet will allow the investigators to avoid inter-individuals variability in making infusion changes standardizing the interventions in two groups.

Actually the traditional system of monitoring of glycemia has been demonstrated to be unable to detect a significant number of glycemic variations during the daytime. Increasing the number of blood glycemic test (by heel prick) would mean to increase the number of painful procedures for the newborn with an uncertain benefit and the workload of the staff.

Disclosures: Dexcom Inc, USA will provide materials for the study as donation to the Neonatal Intensive Care Unit of University Hospital of Padua, Italy.

The study has been designed as a no-profit research project by the Principal Investigators and Collaborators of Neonatal Intensive Care Unit of University of Padua, Department of Bioengineering (University of Padua) and Boston Children's Hospital.

Dexcom Inc has not been involved in the study design and will not be involved in results evaluation.

ELIGIBILITY:
Inclusion Criteria (and/or):

* <= 32 weeks gestation
* birthweight <1500 g

Exclusion Criteria:

* birthweight <500g
* malformative syndrome
* lack of parental consent
* chromosomal abnormalities

Ages: 2 Hours to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
In range - time | 7 days (minimum 2)
  Percentage of time in range 72-144mg/dl

SECONDARY OUTCOMES:
Hypoglycemia | 7days
  percentage of time below 40mg/dl
Acute event associated to glycemic variability and/or hypoglycemia | 7days
  Acute events (cerebral hemorrhage) and association with glycemic variability (specific patterns)
Glycemic variability and hypoglycemia predictors | 7days
  Evaluation of glycemic variability
hypoglycemia prediction | 7days
  Predictors of hypoglycemia: to individuate glycemic patterns/trends that could predict hypoglycemia
Glycemic modeling | 7days
  Creation of a glycemic modeling to predict hypoglycemia and to prevent it (see Klonoff DC et al J Diabetes Sci Technol. 2010)
Pain associated to insertion of CGM respect to Pain associated to heel prick | 7 days
  PIPP scale will be used to compare CGM vs heel prick in each subject. The scale consists of a numeric score as described by Stevens B (Clin J Pain, 1996)

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Galderisi, MD, Principal Investigator — University Hospital of Padua; Daniele Trevisanuto, MD, Principal Investigator — University Hospital of Padua
Locations (3):
- Boston Children's Hospital, Boston, Massachusetts, United States
- Italy (2):
  - Neonatal Intensive Care Unit - University Hospital of Padua, Padua, Padua
  - Department of Information Engineering - University of Padua, Padua, Padua

REFERENCES:
- [Result] Agus MS, Steil GM, Wypij D, Costello JM, Laussen PC, Langer M, Alexander JL, Scoppettuolo LA, Pigula FA, Charpie JR, Ohye RG, Gaies MG; SPECS Study Investigators. Tight glycemic control versus standard care after pediatric cardiac surgery. N Engl J Med. 2012 Sep 27;367(13):1208-19. doi: 10.1056/NEJMoa1206044. Epub 2012 Sep 7. PMID 22957521
- [Result] Beardsall K, Vanhaesebrouck S, Ogilvy-Stuart AL, Vanhole C, Palmer CR, Ong K, vanWeissenbruch M, Midgley P, Thompson M, Thio M, Cornette L, Ossuetta I, Iglesias I, Theyskens C, de Jong M, Gill B, Ahluwalia JS, de Zegher F, Dunger DB. Prevalence and determinants of hyperglycemia in very low birth weight infants: cohort analyses of the NIRTURE study. J Pediatr. 2010 Nov;157(5):715-9.e1-3. doi: 10.1016/j.jpeds.2010.04.032. Epub 2010 Jun 8. PMID 20570286
- [Result] Beardsall K, Vanhaesebrouck S, Ogilvy-Stuart AL, Vanhole C, Palmer CR, van Weissenbruch M, Midgley P, Thompson M, Thio M, Cornette L, Ossuetta I, Iglesias I, Theyskens C, de Jong M, Ahluwalia JS, de Zegher F, Dunger DB. Early insulin therapy in very-low-birth-weight infants. N Engl J Med. 2008 Oct 30;359(18):1873-84. doi: 10.1056/NEJMoa0803725. PMID 18971490
- [Result] Burns CM, Rutherford MA, Boardman JP, Cowan FM. Patterns of cerebral injury and neurodevelopmental outcomes after symptomatic neonatal hypoglycemia. Pediatrics. 2008 Jul;122(1):65-74. doi: 10.1542/peds.2007-2822. PMID 18595988
- [Result] Committee on Fetus and Newborn; Adamkin DH. Postnatal glucose homeostasis in late-preterm and term infants. Pediatrics. 2011 Mar;127(3):575-9. doi: 10.1542/peds.2010-3851. Epub 2011 Feb 28. PMID 21357346
- [Result] Cornblath M, Hawdon JM, Williams AF, Aynsley-Green A, Ward-Platt MP, Schwartz R, Kalhan SC. Controversies regarding definition of neonatal hypoglycemia: suggested operational thresholds. Pediatrics. 2000 May;105(5):1141-5. doi: 10.1542/peds.105.5.1141. PMID 10790476
- [Result] Duvanel CB, Fawer CL, Cotting J, Hohlfeld P, Matthieu JM. Long-term effects of neonatal hypoglycemia on brain growth and psychomotor development in small-for-gestational-age preterm infants. J Pediatr. 1999 Apr;134(4):492-8. doi: 10.1016/s0022-3476(99)70209-x. PMID 10190926
- [Result] Hay WW Jr, Raju TN, Higgins RD, Kalhan SC, Devaskar SU. Knowledge gaps and research needs for understanding and treating neonatal hypoglycemia: workshop report from Eunice Kennedy Shriver National Institute of Child Health and Human Development. J Pediatr. 2009 Nov;155(5):612-7. doi: 10.1016/j.jpeds.2009.06.044. No abstract available. PMID 19840614
- [Result] Wong DS, Poskitt KJ, Chau V, Miller SP, Roland E, Hill A, Tam EW. Brain injury patterns in hypoglycemia in neonatal encephalopathy. AJNR Am J Neuroradiol. 2013 Jul;34(7):1456-61. doi: 10.3174/ajnr.A3423. Epub 2013 Feb 22. PMID 23436054
- [Result] McKinlay CJ, Alsweiler JM, Ansell JM, Anstice NS, Chase JG, Gamble GD, Harris DL, Jacobs RJ, Jiang Y, Paudel N, Signal M, Thompson B, Wouldes TA, Yu TY, Harding JE; CHYLD Study Group. Neonatal Glycemia and Neurodevelopmental Outcomes at 2 Years. N Engl J Med. 2015 Oct 15;373(16):1507-18. doi: 10.1056/NEJMoa1504909. PMID 26465984
- [Result] Stevens B, Johnston C, Petryshen P, Taddio A. Premature Infant Pain Profile: development and initial validation. Clin J Pain. 1996 Mar;12(1):13-22. doi: 10.1097/00002508-199603000-00004. PMID 8722730
- [Result] Klonoff DC. The need for a glycemia modeling comparison workshop to facilitate development of an artificial pancreas. J Diabetes Sci Technol. 2010 Jan 1;4(1):1-3. doi: 10.1177/193229681000400101. No abstract available. PMID 20167161
- [Derived] Galderisi A, Zammataro L, Losiouk E, Lanzola G, Kraemer K, Facchinetti A, Galeazzo B, Favero V, Baraldi E, Cobelli C, Trevisanuto D, Steil GM. Continuous Glucose Monitoring Linked to an Artificial Intelligence Risk Index: Early Footprints of Intraventricular Hemorrhage in Preterm Neonates. Diabetes Technol Ther. 2019 Mar;21(3):146-153. doi: 10.1089/dia.2018.0383. PMID 30835533
- [Derived] Galderisi A, Lago P, Steil GM, Ghirardo M, Cobelli C, Baraldi E, Trevisanuto D. Procedural Pain during Insertion of a Continuous Glucose Monitoring Device in Preterm Infants. J Pediatr. 2018 Sep;200:261-264.e1. doi: 10.1016/j.jpeds.2018.03.040. Epub 2018 May 31. PMID 29861315